CLINICAL TRIAL: NCT05501197
Title: Comparison of the Effects of Different Telerehabilitation Methods on Pain, Functional Limitation, Muscle Strength, Balance, and Quality of Life in Patients With Meniscus Degeneration
Brief Title: Effects of Different Telerehabilitation Methods on Pain, Functional Limitation, Muscle Strength, Balance, and Quality of Life in Patients With Meniscus Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eren Timurtas, PhD, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2022.602/2
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Meniscus; Degeneration
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telerehabilitation Group (Active Comparator): Synchronous Telerehabilitation Group will receive exercise therapy via video conference.
  Interventions: Other: Exercise Therapy via video conference
- Asynchronous Telerehabilitation Group (Experimental): Asynchronous Telerehabilitation Group will receive exercise therapy via mobile application.
  Interventions: Other: Exercise Therapy via mobile application

INTERVENTIONS:
Other: Exercise Therapy via video conference — The intervention will include the different levels of the following exercises that are given to the patient considering their functional level:
  Straight leg raise (Level 1-2-3) Quadriceps strengthening (Level 1-2-3) Hip abductor/adductor strengthening (Level 1-2-3) Hamstring stretch Gastrocnemius stretch
  Other Names: Therapeutic Exercise
  Arms: Synchronous Telerehabilitation Group
Other: Exercise Therapy via mobile application — The intervention will include the different levels of the following exercises that are given to the patient considering their functional level:
  Straight leg raise (Level 1-2-3) Quadriceps strengthening (Level 1-2-3) Hip abductor/adductor strengthening (Level 1-2-3) Hamstring stretch Gastrocnemius stretch
  Other Names: Therapeutic Exercise
  Arms: Asynchronous Telerehabilitation Group

SUMMARY:
Our study will include 60 patients diagnosed with meniscus degeneration in the Department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences of Marmara University. Volunteers will be informed about the purpose of the study and the evaluations and treatments to be carried out, and their consent will be obtained by reading the 'Informed Volunteer Consent Form' and obtaining their signatures. The sample group and distribution will be determined as 30 asynchronous telerehabilitation groups and 30 synchronous telerehabilitation groups. Our study is a randomized controlled trial. Groups will be formed in a randomized manner and blinded study design will be used to evaluate outcome parameters. Patients beginning the rehabilitation program will be evaluated at the start of the study, at week 4, week 8, and week 16. Demographic information of the patients participating in the study will be obtained using the demographic data form. Visual Analogue Scale (VAS) for pain, WOMET index for functionality and quality of life, functionality with Lysholm Knee Scoring Scale and quality of life with Patient Generated Index (PGI) and Short Form-12 (SF-12) scales; Functional mobility Timed Up and Go Test (TUG), functional capacity 2 Minutes Walk Test (2 MWT), balance Balance Master, proprioception and muscle strength Isokinetic assessment device, lower extremity neuromuscular function level 30 sec Sit Up and 5 Sit & Go performance tests will be evaluated with Our study will investigate the comparison of the effects of asynchronous and synchronous telerehabilitation programs on pain, functional limitation, muscle strength and quality of life in patients with meniscal degeneration.

DETAILED DESCRIPTION:
Meniscus degeneration is a common problem in the society and is a health problem that can be seen at any age and affects a large part of the population. The functions of the menisci are load bearing, load transfer, shock absorption and lubrication. Meniscus degeneration occurs as a part of the degenerative process of the knee joint and shows symptoms such as pain and instability in people, and these symptoms are associated with functional limitation. Treatment of meniscus degeneration can be classified as pharmacological, non-pharmacological and surgical treatment. Nonpharmacological treatment uses traditional physiotherapy and rehabilitation approaches such as patient education, exercise therapy, and various physiotherapy applications. Exercises used in the treatment of meniscus degeneration aim to reduce pain, provide joint range of motion, increase knee joint functions, protect muscle strength and joint proprioception. Thus, it is predicted that the participation of patients in social life will increase.

With the developing technology, telerehabilitation applications appear as an alternative approach to traditional physiotherapy approaches. Telerehabilitation provides access to patients by using information and communication technologies and provides rehabilitation services in this way. There are two types of telerehabilitation, synchronous and asynchronous rehabilitation. Applications that allow instant interaction via a webcam for synchronous rehabilitation, telephone or video conferencing connection. Asynchronous rehabilitation, on the other hand, can be defined as applications that transmit recorded video and audio recording data for later interpretation by a specialist. Studies on telerehabilitation are limited in the literature. There are no studies measuring the effectiveness of asynchronous and synchronous telerehabilitation in patients with meniscal degeneration. Especially under the conditions of the COVID-19 pandemic, patients cannot get an appointment for the physiotherapy service, the waiting time for treatment is prolonged, physiotherapy and rehabilitation services are costly, the patients have difficulty in reaching the physiotherapy service due to their geographical location, especially the patients who complain of lower extremity problems travel long distances and reach the rehabilitation unit in long hours. For this reason, the inability to get efficiency from physical therapy enabled us to conduct research on telerehabilitation.

Our study will include 60 patients diagnosed with meniscus degeneration in the Department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences of Marmara University. Volunteers will be informed about the purpose of the study and the evaluations and treatments to be carried out, and their consent will be obtained by reading the 'Informed Volunteer Consent Form' and obtaining their signatures. The sample group and distribution will be determined as 30 asynchronous telerehabilitation groups and 30 synchronous telerehabilitation groups. Our study is a randomized controlled trial. Groups will be formed in a randomized manner and blinded study design will be used to evaluate outcome parameters. Patients beginning the rehabilitation program will be evaluated at the start of the study, at week 4, week 8, and week 16. Demographic information of the patients participating in the study will be obtained using the demographic data form. Visual Analogue Scale (VAS) for pain, WOMET index for functionality and quality of life, functionality with Lysholm Knee Scoring Scale and quality of life with Patient Generated Index (PGI) and Short Form-12 (SF-12) scales; Functional mobility Timed Up and Go Test (TUG), functional capacity 2 Minutes Walk Test (2 MWT), balance Balance Master, proprioception and muscle strength Isokinetic assessment device, lower extremity neuromuscular function level 30 sec Sit Up and 5 Sit & Go performance tests will be evaluated with Our study will investigate the comparison of the effects of asynchronous and synchronous telerehabilitation programs on pain, functional limitation, muscle strength and quality of life in patients with meniscal degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Pain less than or equal to 7 according to VAS
* Individuals aged 18-65
* Patients with independent mobility

Exclusion Criteria:

* Patients who have undergone surgery in the last 1 year
* Patients who have undergone total knee replacement or total hip replacement surgery
* Patients with acute trauma in the last 1 year
* Patients with uncontrolled chronic disease
* Patients who have received physical therapy in the last 6 months
* Patients who have received hyaluronic acid and corticosteroid injections in the last 6 months
* Patients with a respiratory condition that interferes with walking will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-08 (Estimated); Primary Completion 2022-12-27 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
The Lysholm score | The The Lysholm score will be measured at baseline 2 minutes after pain assessment.
  The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting.
The Lysholm score | The The Lysholm score will be measured at the end of intervention (8. week) 2 minutes after pain assessment.
  The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting.
Visual analogue scale (VAS) | The pain will be measured at baseline
  Pain will be measured using a 10 cm visual analogue scale (VAS). The participants places a mark on the line that best represented their perception of pain at that instant. The VAS score will be measured in cm from the left hand end of the line to the mark.
Visual analogue scale (VAS) | The pain will be measured at the end of intervention (8. week).
  Pain will be measured using a 10 cm visual analogue scale (VAS). The participants places a mark on the line that best represented their perception of pain at that instant. The VAS score will be measured in cm from the left hand end of the line to the mark.

SECONDARY OUTCOMES:
12-Item Short Form Survey (SF-12) | The SF-12 will be measured at baseline 2 minutes after The Lysholm score assessment.
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. The SF-12 was created to reduce the burden of response.
  The SF-12 uses the same eight domains as the SF-36:
  Limitations in physical activities because of health problems. Limitations in social activities because of physical or emotional problems Limitations in usual role activities because of physical health problems Bodily pain General mental health (psychological distress and well-being) Limitations in usual role activities because of emotional problems Vitality (energy and fatigue) General health perceptions
12-Item Short Form Survey (SF-12) | The SF-12 will be measured at the end of intervention (8. week) 2 minutes after The Lysholm score assessment.
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. The SF-12 was created to reduce the burden of response.
  The SF-12 uses the same eight domains as the SF-36:
  Limitations in physical activities because of health problems. Limitations in social activities because of physical or emotional problems Limitations in usual role activities because of physical health problems Bodily pain General mental health (psychological distress and well-being) Limitations in usual role activities because of emotional problems Vitality (energy and fatigue) General health perceptions
30 Seconds Sit To Stand Test | The 30 Seconds Sit To Stand Test will be measured at baseline 2 minutes after SF-12 assessment.
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults. The 30-Second Chair Test is administered using a folding chair without arms, with seat height of 17 inches (43.2 cm). The chair, with rubber tips on the legs, is placed against a wall to prevent it from moving.
  The participant is seated in the middle of the chair, back straight; feet approximately a shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest.
  Have the patient practice a repetition or two before completing the test. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.
30 Seconds Sit To Stand Test | The 30 Seconds Sit To Stand Test will be measured at the end of intervention (8. week) 2 minutes after SF-12 assessment.
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults. The 30-Second Chair Test is administered using a folding chair without arms, with seat height of 17 inches (43.2 cm). The chair, with rubber tips on the legs, is placed against a wall to prevent it from moving.
  The participant is seated in the middle of the chair, back straight; feet approximately a shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest.
  Have the patient practice a repetition or two before completing the test. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.
2 Minute Walk Test | The 2 Minute Walk Test will be measured at baseline 5 minutes after 30 Seconds Sit To Stand Test assessment.
  The Two/2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity.
  The person is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured.
  Start timing when the individual is instructed to "Go". Stop timing at 2 minutes. Assistive devices can be used but should be kept consistent and documented from test to test.
  If physical assistance is required to walk, the test should not be performed. The measuring wheel is helpful to determine the distance walked. The person should walk at the fastest speed possible. Rest breaks are allowed if needed.
  Before starting the test, the observer gives initial instructions.
2 Minute Walk Test | The 2 Minute Walk Test will be measured at the end of intervention (8. week) 5 minutes after 30 Seconds Sit To Stand Test assessment.
  The Two/2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity.
  The person is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured.
  Start timing when the individual is instructed to "Go". Stop timing at 2 minutes. Assistive devices can be used but should be kept consistent and documented from test to test.
  If physical assistance is required to walk, the test should not be performed. The measuring wheel is helpful to determine the distance walked. The person should walk at the fastest speed possible. Rest breaks are allowed if needed.
  Before starting the test, the observer gives initial instructions.
Quadriceps and Hamstring Muscle Strength | The Quadriceps and Hamstring Muscle Strength will be measured at baseline 15 minutes after 2 Minute Walk Test assessment.
  Isometric muscle strength of the Quadriceps Femoris and Hamstring muscle groups will be measured at 30º and 60º using the Biodex® System Pro3 (Biodex Corp. Shirley NY, USA) isokinetic test dynamometer. During the test, the back angle of the dynamometer seat is adjusted to 85° and the patients are asked to hold on to the bars next to the seat. The leg to be tested is fixed with the help of belts to prevent compensation of the pelvis and trunk. The test protocol was explained to the patients beforehand; They were instructed to apply force (30º and 60º angle) to the specified area of the device with as much effort as they could and not to allow the device to move their extremities. Before the isometric muscle strength test is performed on the isokinetic system, the patients were given 3 repetitive exercises. The dynamometric test was first performed with 3 repetitions at an angle of 30º, and then 3 repetitions at 60º. 15 seconds between tests, rest periods are given.
Quadriceps and Hamstring Muscle Strength | The Quadriceps and Hamstring Muscle Strength will be measured at the end of intervention (8. week) 15 minutes after 2 Minute Walk Test assessment.
  Isometric muscle strength of the Quadriceps Femoris and Hamstring muscle groups will be measured at 30º and 60º using the Biodex® System Pro3 (Biodex Corp. Shirley NY, USA) isokinetic test dynamometer. During the test, the back angle of the dynamometer seat is adjusted to 85° and the patients are asked to hold on to the bars next to the seat. The leg to be tested is fixed with the help of belts to prevent compensation of the pelvis and trunk. The test protocol was explained to the patients beforehand; They were instructed to apply force (30º and 60º angle) to the specified area of the device with as much effort as they could and not to allow the device to move their extremities. Before the isometric muscle strength test is performed on the isokinetic system, the patients were given 3 repetitive exercises. The dynamometric test was first performed with 3 repetitions at an angle of 30º, and then 3 repetitions at 60º. 15 seconds between tests, rest periods are given.

IPD SHARING:
Plan to Share IPD: No